CLINICAL TRIAL: NCT06765187
Title: Cross-sectional Study to Assess Tolerability of the Trivalent Recombinant Vaccine in Individuals Between 18 and 64 Years Old Using the Vaccinees Perception of Injection.
Status: Completed | Type: Observational
Sponsor: Sanofi Pasteur, a Sanofi Company (Industry)
Responsible Party: Sponsor
Organization: Sanofi (Industry)
Other Study IDs: VAP00035
Record Dates: First submitted 2024-12-18; First posted 2025-01-09 (Actual); Last update posted 2025-02-13 (Actual); Status verified 2025-02

CONDITIONS: Influenza Immunization; Health Volunteers
MeSH Terms: conditions — Influenza, Human

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes

GROUPS / COHORTS (1):
- Group 1: Individuals who have received flu vaccine RIV3 within 2 months prior to being contacted
  Interventions: Biological: RIV3

INTERVENTIONS:
Biological: RIV3 — intramuscular injection

SUMMARY:
This study aims to assess patient-reported experiences post-vaccination with RIV3 using the VAPI instrument, identify drivers for vaccine choice in each case, and assess the cross-validity of VAPI, by establishing magnitude of correlations to EQ-5D-5L domains.

As a feasibility endpoint, this study aims to describe the socio-demographic differences and feasibility of matching between recipients of RIV3 vaccine and mRNA vaccines for COVID-19.

DETAILED DESCRIPTION:
This study will be conducted through an online survey that respondents will complete only if they meet the inclusion criteria and give their consent to continue to the main questionnaire. Each participant will complete the survey only once. Participants will provide details about their demographic data, health status, perceptions of flu vaccination and injection site reactions, as well as drivers for vaccine choice and future vaccine use.

ELIGIBILITY:
Inclusion Criteria:

* Be aged 18-64 years old
* 50 to 64 years will be the main age group for recruitment
* 18 to 49 years will allow flexibility to face potential recruitment challenges
* Have received a RIV3 vaccine within the last 2 months
* Be able to provide explicit consent to participate in the study
* Reside in continental US (Puerto Rico is excluded)
* Communicate and read fluently in English (US)
* Be physically able to participate in a 30 min online survey using an internet-enabled computer or other device (such as a tablet or smartphone)

Exclusion Criteria:

* Inability to participate in survey
* Receipt of any other vaccine outside those pre-specified within the past three weeks, and including concomitant vaccination
* Receipt of co-administered vaccination

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Vaccine recipients who meet the inclusion criteria will be recruited from the United States of America (USA) over a period of 3 to 4 months. The study will include a sample of vaccine recipients, called group 1, and will recruit individuals who have received flu vaccine RIV3.
Sampling Method: Probability Sample
Enrollment: 447 (Actual)
Dates: Start 2024-11-18 (Actual); Primary Completion 2025-01-04 (Actual); Study Completion 2025-01-04 (Actual)

PRIMARY OUTCOMES:
Incidence of reactions (local) | At the time of inclusion in the study
  Vaccinees' Perception of Injection (VAPI) and EQ-5D-5L questionnaires will be used. VAPI questionnaire consists of four dimensions. The first dimension collects information on discomfort caused by reactions at the injection site. The second dimension covers local reactions. The third dimension gathers data on pain. The fourth dimension collects information on acceptability and intentions for vaccination in the next year. The EQ-5D-5L instrument consists of two main components. The first part includes five dimensions of health: Mobility, Self-care, Usual activities, Pain/discomfort, and Anxiety/depression. The second part comprises a vertical scale where respondents rate their overall health. The higher the score the worse is the experience.
Incidence of reactions (systemic) | At the time of inclusion in the study
  Vaccinees' Perception of Injection (VAPI) and EQ-5D-5L questionnaires will be used. VAPI questionnaire consists of four dimensions. The first dimension collects information on discomfort caused by reactions at the injection site. The second dimension covers local reactions. The third dimension gathers data on pain. The fourth dimension collects information on acceptability and intentions for vaccination in the next year. The EQ-5D-5L instrument consists of two main components. The first part includes five dimensions of health: Mobility, Self-care, Usual activities, Pain/discomfort, and Anxiety/depression. The second part comprises a vertical scale where respondents rate their overall health. The higher the score the worse is the experience.
Severity of reactions (local and systemic) | At the time of inclusion in the study
  Vaccinees' Perception of Injection (VAPI) and EQ-5D-5L questionnaires will be used. VAPI questionnaire consists of four dimensions. The first dimension collects information on discomfort caused by reactions at the injection site. The second dimension covers local reactions. The third dimension gathers data on pain. The fourth dimension collects information on acceptability and intentions for vaccination in the next year. The EQ-5D-5L instrument consists of two main components. The first part includes five dimensions of health: Mobility, Self-care, Usual activities, Pain/discomfort, and Anxiety/depression. The second part comprises a vertical scale where respondents rate their overall health. The higher the score the worse is the experience.
vaccine acceptability score | At the time of inclusion in the study
  VAPI and EQ-5D-5L questionnaires will be used.
impact on daily life activities score | At the time of inclusion in the study
  VAPI and EQ-5D-5L questionnaires will be used.

SECONDARY OUTCOMES:
Frequencies of factors driving patient choices of RIV3 score | At the time of inclusion in the study
  VAPI and EQ-5D-5L questionnaires will be used.
Proportions of factors driving patient choices of RIV3 score | At the time of inclusion in the study
  VAPI and EQ-5D-5L questionnaires will be used.
Correlation score between EQ-5D-5L and VAPI questionaries | At the time of inclusion in the study
  By examining the correlation between these domains, the study intends to better understand how perceptions of injection-related adverse effects corelate to broader measures of health-related quality of life, notably those coming from a gold-standard and simpler instrument

CONTACTS AND LOCATIONS:
Locations (1):
- Investigational site, Swiftwater, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to patient level data and related study documents including the clinical study report, study protocol with any amendments, blank case report form, statistical analysis plan, and dataset specifications. Patient level data will be anonymized and study documents will be redacted to protect the privacy of trial participants. Further details on Sanofi's data sharing criteria, eligible studies, and process for requesting access can be found at: https://vivli.org